CLINICAL TRIAL: NCT06610838
Title: Longitudinal Effects of E-cigarette Use on Cardiovascular and Pulmonary Health
Brief Title: Effects of E-cigarette Use on Health
Acronym: VAPECHECK
Status: Recruiting | Type: Observational
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 2024-0684; 1R01HL175602-01 (NIH); A534253 (Other: UW- Madison); SMPH/MEDICINE/GEN INT MD (Other: UW- Madison); Protocol Version 10/23/25 (Other: UW Madison)
Record Dates: First submitted 2024-09-19; First posted 2024-09-24 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Electronic Cigarette Use
MeSH Terms: conditions — Vaping

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ENDS users: Long-term stable users of electronic nicotine delivery systems, 21 years of age or older, who do not use combustible (conventional) cigarettes
  Interventions: Other: Health Assessments
- Non-users: Gender-matched control participants who do not use ENDS or combustible cigarettes
  Interventions: Other: Health Assessments

INTERVENTIONS:
Other: Health Assessments — Participants will complete the blood tests, questionnaires, cardiovascular tests, and pulmonary test at visits 1, 2, and 4. Non-Contrast Chest CT and cardiopulmonary treadmill (VO2 max) stress tests will occur at visits 1 and 4. Visit 3 will not include cardiovascular and pulmonary tests.

SUMMARY:
Electronic nicotine delivery systems (ENDS) are used by millions of Americans, however their long-term health effects are unknown. This research proposal will quantify the effects of long-term ENDS use on validated and novel biomarkers of cardiovascular and pulmonary disease and how they are influenced by use heaviness, age, body weight, and co-use of other products. This study will produce the most informative evidence to date on how long-term ENDS use affects cardiovascular and pulmonary health.

DETAILED DESCRIPTION:
Electronic nicotine delivery systems (ENDS) are used by millions of Americans, however, their long-term health effects are unknown. Although ENDS use delivers far lower levels of carcinogens than tobacco smoking, very little is known about whether ENDS use affects the risks of developing cardiovascular (CV) or pulmonary diseases, two of the most highly prevalent causes of morbidity and mortality in the United States. This research proposal will quantify the effects of long-term ENDS use on validated and novel biomarkers of CV and pulmonary disease and how they are influenced by use heaviness, age, body weight, and co-use of other products. This research also will shed additional light on long-term ENDS use patterns and ENDS dependence. The importance of this study does not rest upon demonstrating adverse effects of ENDS use.

The study team will recruit up to 400 long-term, stable users of ENDS and up to 200 age- and gender-matched control participants who do not use ENDS or combustible cigarettes. They will undergo comprehensive biomarker assessments over 36 months. Biomarkers assess CV and pulmonary health status and risk and include vital signs, blood samples for systemic inflammation and oxidative stress, lipids, and markers of insulin resistance and cardiometabolic health. Arterial structure changes will be assessed using carotid ultrasound. Sympathetic nervous system activation will be assessed by heart rate variability and arterial diameters. For pulmonary measures, the study team will obtain non-contrast quantitative computed tomography (CT) images to assess air trapping and texture-based measures of inflammation. The researcher also will perform spirometry. Integrated cardiopulmonary health will be assessed via treadmill stress testing. Other measures will include exhaled carbon monoxide, real-time measures of nicotine product use, nicotine dependence, and use of cannabis and alcohol. Biomarker status over time will be compared across groups and related to ENDS use heaviness, use of other products, and person factors (i.e., age, gender, race/ethnicity, weight, and smoking history). About 130 participants who were phenotyped from 2019-2021 will be included.

The Primary Aim is to determine relationships between ENDS use heaviness and changes in our CV and pulmonary health biomarkers over 3 years. Biomarker status across ENDS users and non-users over time will be compared and associations between biomarker status and ENDS use heaviness within the ENDS user group will be examined.

The Secondary Aim is to characterize changes in ENDS use patterns and dependence over time and to determine how these are related to biomarker status changes and how they are influenced by the person factors described above. The primary and secondary CV measures are changes in common carotid artery intima-media thickness (CCA IMT) and grayscale median (GSM). The primary and secondary pulmonary measures are the changes in the quantitative CT measures of air trapping and parenchymal texture. This proposal will produce the most informative evidence to date on how long-term ENDS use affects CV and pulmonary health and disease risk.

ELIGIBILITY:
Inclusion Criteria:

* greater than or equal to 21 years of age
* has vaped a nicotine e-cigarette product at least 2 days/week for most weeks for greater than or equal to 12 months
* plans to remain in catchment area for greater than or equal to 3 years
* smoked 5 or fewer tobacco cigarettes in the past 6 months
* no serious CV, pulmonary, or other medical problems
* not currently pregnant
* no plans to stop vaping

Exclusion Criteria:

* serious CV, pulmonary, or other medical problems (e.g., moderate or severe aortic stenosis, class III or IV heart failure, blood pressure greater than or equal to 160/100 mmHg, interstitial lung disease, sarcoidosis, Stage 3 or 4 cancer)
* combusted or vaped cannabis use 3 days/week or more in the past 3 months
* currently pregnant
* not able to read an write English
* incarceration

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The participants enrolled will comprise a large group of exclusive ENDS users who do not use combusted cigarettes and who have used ENDS regularly for at least 1 year. ENDS participants must have vaped at least 2 days/week for greater than or equal to 12 months, smoke very infrequently, and have no plans to try to stop vaping in the foreseeable future. The comparison non-user group also will be gender-matched and comprise those who report no vaping or smoking in the past 6 months and less than 5 times in 2 years.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2025-01-06 (Actual); Primary Completion 2029-06-30 (Estimated); Study Completion 2029-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in mean common carotid artery intima-media thickness (CCA-IMT) | Baseline to 3 years
  Carotid ultrasound CCA-IMT measures the thickness of the carotid artery wall and is a measure of arterial injury. Rates of change vary by age, sex, and race, but less increase is associated with less cardiovascular disease risk.
Change in LAA-856 | Baseline to 3 years
  Quantitative computed tomography (CT) can measure LAA-856 [percent of lung voxels less than -856 HU], which describes air trapping. Less air trapping indicates less progression of obstructive ventilation in and risk of obstructive lung diseases.

SECONDARY OUTCOMES:
Change in common carotid artery intima-media Grayscale Median (GSM) | Baseline to 3 years
  Changes in Parenchymal Texture will be in part measured with carotid GSM. Captured via ultrasound, images analyzed using LifeQ Medical Plaque Analysis Software for GSM.

CONTACTS AND LOCATIONS:
Overall Officials: Timothy Baker, PhD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- UW Center for Tobacco Research and Intervention, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: Yes
All of the questionnaire and interview responses, the ecological momentary assessment (EMA) data, results of cardiovascular and pulmonary tests, and urine and blood test results will be preserved and shared to the Biologic Specimen and Data Repository (BioLINCC) in comma separated value (CSV) format.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: The study team will submit processed and cleaned data to the Biologic Specimen and Data Repository (BioLINCC) approximately 3 months prior to any publication date or 3 months after the end of the performance period, whichever is sooner. Data will be available indefinitely (i.e., for as long as the BioLINCC repository is maintained or chooses to continue to archive our study data).
Access Criteria: Data will be shared with controlled access in BioLINCC for general research use, as allowed by the participant's informed consent agreement and the Institutional Certification.